CLINICAL TRIAL: NCT00699400
Title: A Phase IV, Prospective, Multicenter, Observational Oocyte Cryopreservation Registry
Brief Title: Oocyte Cryopreservation Registry (HOPE Registry)
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: 28599
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Oocyte Cryopreservation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Phase IV, prospective multicenter, observational Registry will track cycle outcomes for subjects who are thawing frozen oocytes for subsequent use through in vitro fertilization (IVF) and embryo transfer (ET)

DETAILED DESCRIPTION:
Subjects will be enrolled at as many ART clinics that offer oocyte cryopreservation and are willing to participate in the Registry. Oocytes will be retrieved and cryopreserved from autologous or heterologous donors. When the subject decides she would like to get pregnant, oocytes will be thawed, fertilized and the resultant embryos will be transferred to the oocyte donor (for autologous use) or to another recipient (for heterologous use). The treatment regimen will be completed with births and well-baby follow-up of children at 12 months of age. Information on children will be submitted by their parents to the Investigators. Data collection for the Registry will be active for a maximum of five (5) years, including three (3) years of enrollment and two (2) additional years to complete the well-baby follow-up for all the children.

ELIGIBILITY:
Inclusion Criteria:

* Must be in an ART program
* Donor and recipients must be of reproductive age (18-50 years old, inclusive at the time of oocyte freezing and/or thawing) who intend to achieve a pregnancy by utilizing frozen thawed autologous or heterologous oocytes
* Female and partner (if applicable) must voluntarily provide written informed consent/HIPAA authorization prior to any Registry-related data collection
* Female and partner (if applicable) must be willing to provide a second written informed consent following each live birth prior to any Registry- related data collection on birth characteristics and twelve (12) month evaluation of offspring
* Children born from women who take part in this registry from birth to 12 months (+/- 1 month) of age

Exclusion Criteria:

* Have clinically significant systemic disease
* Have abnormal, undiagnosed gynecological bleeding
* Have any contraindication to Controlled Ovarian Stimulation (COS) for ART and to gonadotropins to be used in ART
* Also, in a rare situation, are undergoing ET with mixed embryos generated from fresh oocytes produced in the current cycle as well as frozen embryos generated from nonfrozen oocytes obtained in a previous ART cycle
* Children born from women who do not take part in this Registry
* Any offspring of woman who are not Registry subjects cannot take part in this registry

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of reproductive age who, in order to achieve a pregnancy, will have embryos created from thawed autologously or heterologously implanted oocytes that were either:
  * cryopreserved at the time of or following the Registry's launch, or
  * cryopreserved prior to the Registry's launch, but will undergo thaw/fertilization/transfer procedures while the subject is enrolled in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mahony, PhD, HCLD (AAB), Study Director — EMD Serono
Locations (14):
- United States (14):
  - Research Site, Fountain Valley, California
  - Research Site, Laguna Hills, California
  - Research Site, Newport Beach, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Glenville, Illinois
  - US Local Med Info Office, Rockland, Massachusetts
  - Research Site, Waltham, Massachusetts
  - Research Site, Millburn, New Jersey
  - Research Stie, New York, New York
  - Research Site, Bryn Mawr, Pennsylvania

REFERENCES:
- [Derived] Nagy ZP, Anderson RE, Feinberg EC, Hayward B, Mahony MC. The Human Oocyte Preservation Experience (HOPE) Registry: evaluation of cryopreservation techniques and oocyte source on outcomes. Reprod Biol Endocrinol. 2017 Feb 7;15(1):10. doi: 10.1186/s12958-017-0228-7. PMID 28173814

RESULTS

PARTICIPANT FLOW:
Groups:
- Slow Freeze (One Cycle): Subjects who participated in one freezing cycle of the Registry only using the slow freeze technique (i.e. freezing that occurs at a slow rate to minimize ice formation)
- Slow Freeze (Two Cycles): Subjects who participated in two freezing cycles of the Registry only using the slow freeze technique (i.e. freezing that occurs at a slow rate to minimize ice formation)
- Vitrification (One Cycle): Subjects who participated in one freezing cycle of the Registry only using the vitrification technique (i.e. cryopreservation using high initial concentrations of cryoprotectant and ultra rapid cooling to solidify the cell without the formation of ice)
- Vitrification (Two Cycles): Subjects who participated in two freezing cycles of the Registry only using the vitrification technique (i.e. cryopreservation using high initial concentrations of cryoprotectant and ultra rapid cooling to solidify the cell without the formation of ice)
- Both (Slow Freeze and Vitrification): Participants who underwent both slow freezing and vitrification cycles (one cycle of each freezing technique).
- Pre-freeze Discontinuations: Participants who enrolled in the study but withdrew before oocyte retrieval or for whom oocyte retrieval failed (had no oocytes to freeze).
Period: Overall Study
Arm/Group | Slow Freeze (One Cycle) | Slow Freeze (Two Cycles) | Vitrification (One Cycle) | Vitrification (Two Cycles) | Both (Slow Freeze and Vitrification) | Pre-freeze Discontinuations
Started | 42 | 3 | 138 | 6 | 4 | 11
Completed | 42 | 3 | 138 | 6 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Population: Subjects were analyzed based on the freeze cycle(s) that were used, therefore, the 4 subjects that used both types of cryopreservation techniques are summarized in both the slow freeze and vitrification arms. These 4 subjects will be double-counted in the "Total (calculated)" column.
Groups:
- Slow Freeze: Subjects that participated in one or more slow-freeze cycles
- Vitrification: Subjects that participated in one or more vitrification cycles
- Total: Total of all reporting groups
Arm/Group | Slow Freeze | Vitrification | Pre-Freeze Discontinuations | Total
Number analyzed (Participants) | 49 | 148 | 11 | 208
Age, Customized [Number; unit: Participants] — Four subjects underwent cryopreservation cycles for both slow-freezing and vitrification
  11 Participants who enrolled in the study but withdrew before oocyte retrieval or for whom oocyte retrieval failed (had no oocytes to freeze) are captured in the Pre-Freeze Discontinuation Arm.
  Participants
    <35 years | 4 | 34 | 5 | 43
    35-37 years | 3 | 24 | 2 | 29
    38-40 years | 15 | 30 | 2 | 47
    41-42 years | 4 | 26 | 0 | 30
    43-44 years | 13 | 15 | 1 | 29
    > 44 years | 10 | 19 | 1 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 148 | 11 | 208
  Male | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 24.6 (5.2) | 23.4 (3.6) | 19.7 (0) | 23.7 (4.1)
Donor Age [Mean (Standard Deviation); unit: Years] | 25.1 (2.7) | 26.0 (2.8) | NA (NA) — Values not available for Pre-freeze Discontinuation Arm. These participants withdrew before oocyte retrieval or the oocyte retrieval procedure failed (had no oocytes to freeze from themselves or from donors). | 25.7 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Thawing Cycle Level Live Birth Rate
Description: Live birth rate per thawing cycle was calculated from the number of live births divided by the number of oocytes thawed less the number of embryos cryopreserved from thawed oocytes, averaged over all thawing cycles.
Time Frame: Birth of one or more live babies
Population: Live birth rate per thaw cycle(%)
Measure: Mean (95% Confidence Interval); unit: % of oocytes thawed per cycle
Units Other Than Participants: Thawing Cycles
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Thawing Cycles) | 54 | 155 | 209
% of oocytes thawed per cycle | 12.4 [7.7 to 20.0] | 15.0 [12.1 to 18.6] | 13.6 [10.5 to 17.7]

2. Secondary Outcome: Oocyte Level Live Birth Rate
Description: Oocyte Level Live Birth Rate was calculated from the total number of live births divided by the total number of oocytes thawed less the total number of embryos cryopreserved from thawed oocytes
Time Frame: Birth of one or more live babies
Measure: Number; unit: % of all oocytes thawed
Units Other Than Participants: Thawed Oocytes - Cryopreserved Embryos
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Thawed Oocytes - Cryopreserved Embryos) | 409 | 1133 | 1542
% of all oocytes thawed | 4.2 | 7.4 | 6.5

3. Secondary Outcome: Number of Live Babies
Time Frame: Birth of one or more live babies
Measure: Number; unit: Number of live births
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number of live births | 17 | 84 | 101

4. Secondary Outcome: Number of Oocytes Frozen
Time Frame: At cryopreservation
Measure: Number; unit: Number of Oocytes Frozen
Units Other Than Participants: Freezing Cycles
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Freezing Cycles) | 52 | 154 | 206
Number of Oocytes Frozen | 1144 | 3721 | 4865

5. Secondary Outcome: Number of Oocytes Thawed
Time Frame: At start of thawing cycle
Measure: Number; unit: Number of oocytes thawed
Units Other Than Participants: Thawing Cycles
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Thawing Cycles) | 54 | 155 | 209
Number of oocytes thawed | 416 | 1282 | 1698

6. Secondary Outcome: Oocyte Survival Rate
Description: Number of oocytes fertilized divided by number of oocytes thawed per thawing cycle
Time Frame: At time of fertilization
Measure: Mean (Standard Deviation); unit: Oocyte survival rate (%)
Units Other Than Participants: Thawing cycles
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Thawing cycles) | 54 | 155 | 209
Oocyte survival rate (%) | 73.2 (26.2) | 83.3 (20.9) | 80.6 (22.8)

7. Secondary Outcome: Implantation Rate
Description: Implantation rate was calculated as the number of fetal sacs per transferred embryo averaged over all thawing cycles
Time Frame: At time of ultrasound after embryo transfer
Measure: Mean (Standard Deviation); unit: Implantation Rate (%)
Units Other Than Participants: Thawing Cycles
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Thawing Cycles) | 54 | 155 | 209
Implantation Rate (%) | 15.9 (24.1) | 41.7 (43.4) | 35.1 (40.9)

8. Secondary Outcome: Number of Clinical Pregnancies
Description: Number of clinical pregnancies defined as the presence of one or more fetal sacs with a heartbeat.
Time Frame: At time of ultrasound after embryo transfer
Population: Participants could have multiple thawing cycles that could lead to multiple embryo transfers. Only successful thaws lead to embryo transfers and only successful embryo transfers lead to clinical pregnancies.
Measure: Number; unit: Number of Clinical Pregnancies
Units Other Than Participants: Embryo Transfers
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Embryo Transfers) | 40 | 119 | 159
Number of Clinical Pregnancies | 18 | 73 | 91

9. Secondary Outcome: Number of Miscarriages
Description: Number of pregnancy outcomes reported as spontaneous abortions
Time Frame: Anytime after embryo transfer
Population: as for outcome 8
Measure: Number; unit: Number of Miscarriages
Units Other Than Participants: Embryo Transfers
Arm/Group | Slow Freezing | Vitrification | All Participants
Number analyzed (Participants) | 49 | 148 | 193
Number analyzed (Embryo Transfers) | 40 | 119 | 159
Number of Miscarriages | 4 | 10 | 14

ADVERSE EVENTS:
Description: Adverse events were not collected during the study. No deaths occurred during the course of the study
Arm/Group | Slow Freezing | Vitrification | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator may disclose confidential information to the extent required by law or court order, provided that they promptly provide to EMD Serono prior notice of such disclosure and provide assistance in obtaining an order protecting Confidential Information from public disclosure.